CLINICAL TRIAL: NCT00908206
Title: A Placebo-controlled, Single-blind, Cross-over, Randomised, fMRI Study Comparing Cue-induced Brain Activation Patterns After a Single Oral Dose of GSK598809 or Placebo in Abstinent Alcoholic Subjects
Brief Title: Effects of GSK598809 on Brain Activation in Abstinent Alcoholics
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study not approved by BfARM
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 109709
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Substance Dependence; Alcohol Dependence
Keywords: Alcoholism; Craving; Dependence; Alcohol
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): Placebo to match GSK598809.
  Interventions: Drug: GSK598809

INTERVENTIONS:
Drug: GSK598809 — Subjects will receive a single 175 mg oral dose of GSK598809.

SUMMARY:
This study will compare the effects of GSK598809 and placebo in alcohol dependent volunteers. A placebo is a pill with no drug in it (i.e. dummy drug) but it is made to look exactly like the real drug.

Subjects will be given one dose of GSK598809 during one visit and placebo during the other visit. These dosing visits will be at least 1 week apart. The study is randomised, which means that a computer programme will decide by chance (like tossing a coin), the order in which subjects will receive GSK598809 or the placebo, or in other words, whether they will receive GSK598809 or placebo first.

The study is blinded, which means the subjects will not know whether they are receiving study drug or placebo first and neither will the doctors at the institute. If necessary for reasons of safety, the study staff can find out exactly what the subject has received.

The study will last for approximately 4 weeks but could be up to 6 weeks, depending on length of time between screening and dosing. From screening the subjects will be alcohol-abstinent, they may be put on medication for treatment of withdrawal symptoms and then will have at least 7 days without any medication before beginning the study medication. During the study the subjects will be inpatients at the Central Institute of Mental Health. All subjects will be required to fill out questionnaires, perform behavioural tasks and undergo MRI and functional MRI (fMRI) scans.

DETAILED DESCRIPTION:
This is a randomised, placebo controlled, cross-over, single-blind study of the effects of GSK598809 (175 mg, single dose) on multiple pharmacodynamic measures assessed by fMRI and rating scales. In one period subjects will receive GSK598809 and in the other, placebo.

Investigator, subject and all staff at site involved with the study will remain blinded throughout the study. The GSK team will be unblinded to the randomisation code. GSK has classed this as a single blind study however as both investigator and subject are blinded it is referred to as double blind in the study design.

Twenty four recently detoxified and not currently on medication, alcohol-dependent subjects on a specialised addiction ward will be the study group. These subjects will be recruited into this study while participating in a intramural treatment program, outside of the protocol. Subjects will remain in the unit for the duration of the study.

Alcohol-dependent subjects who enter the institutes' treatment program will be screened between 28 and 15 days prior to the first dose of the study medication according to the eligibility criteria. Subjects who satisfy the inclusion and exclusion criteria will be entered into the study. Along with the study procedures described within this protocol, subjects will participate in the institutes standardized inpatient behavioral addiction treatment program outside of the protocol.

Alcohol-dependent participants have to fulfil diagnostic criteria of alcohol dependence as detailed in the eligibility criteria. The severity of alcoholism will be assessed with the Alcohol Dependence Scale and the amount of lifetime alcohol intake will be measured with Lifetime Drinking History.

After the final alcoholic drink and prior to the first dose of study medication subjects will be treated with detoxification medication (lorazepam) for withdrawal symptoms for up to seven days. Following the treatment of withdrawal symptoms, subjects will have a medication free period for at least seven days to ensure the detoxification medication has been washed out. Liver function tests will be performed again at Day -1 of each dosing day and must be in line with criteria.

Subjects will be randomised to one of two sequence: Placebo received first followed by GSK598809, or GKS598809 received first followed by Placebo. Between 8 and 14 days after the last dose of withdrawal medication, subjects will have their first dose of study medication and first MRI scan. At least 7 days and less than 10 days after the first dose/scanning day subjects will receive their second dosing and their second MRI scan.

All subjects will undergo the following battery of minimal risk procedures during the study; filling out questionnaires, performing agreed behavioural tasks, scanning procedures including fMRI and structural MRI (baseline). Alcohol abstinence will be confirmed by random alcohol-breath tests.

Craving for alcohol will be measured with the Alcohol Urge Questionnaire (AUQ) and the Obsessive Compulsive Drinking Scale (OCDS) before each fMRI scanning session and the Alcohol Craving Questionnaire before and after each fMRI scanning session. Nicotine consumption will be assessed with the Fagerstrom Test for nicotine dependence both at screening and on the day prior to each dosing day.

As described above subjects will undergo two MRI scanning sessions of about 1h (1.5h maximum) each, at intervals of at least one week. The scanning will take place after the administration of study medication (GSK598809 or placebo). The single dose of GSK598809 or placebo will be administered about 1-2 h prior to the scan.

The MRI scanning session will start with acquisition of structural MRI brain images to be used as an anatomical reference. The acquisition of the structural MRI will last for around 6 minutes and during this time subjects are able to get familiar with the MRI procedure. Fear and arousal will decline slowly after the first minutes and prior to the fMRI paradigms. Three fMRI paradigms have been selected to probe reactivity to alcohol-related cues, monetary reward, and to measure BOLD signal fluctuations in the brain resting state. Subjects will be discharged from the inpatient unit 2 days (48 hours) after the second fMRI scan; they will be motivated to remain abstinent and returned to their previous living situation.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependent for at least 2 years.
* Willing to use appropriate contraception method.
* Weight less than 120 kg.
* BMI within the range 18.5 - 33 kg/m2.

Exclusion Criteria:

* Heavy smokers (more than 25 cigarettes per day).
* Liver cirrhosis.
* Pregnant or breast feeding female.
* Psychiatric disorder.
* Substance dependence or abuse other than alcoholism and nicotine dependence.
* Medical illness.
* ECG abnormality (personal or family history).
* Sudden unexplained death or syncope in first degree relative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
BOLD signal changes in the relevant brain areas following presentation of visual alcohol-related vs neutral, non-alcohol related cues. | 1.5h (± 0.5h) after each dose (2 doses)
BOLD signal changes in the same brain structures and circuits as above during a Monetary Incentive Delay task. | 1.5h (± 0.5h) after each dose (2 doses)

SECONDARY OUTCOMES:
Subjective craving in response to alcohol-related cues measured with the Alcohol Urge Questionnaire (AUQ) and the Obsessive Compulsive Drinking Scale (OCDS). | Screening and pre-scan.
Spontaneously reported adverse events, laboratory values, cardiovascular variables (blood pressure, heart rate, and ECG variables), temperature, respiratory rate, serum prolactin concentrations, TSH, testosterone, LH and FSH. | Throughout study.
Pharmacokinetic parameters of GSK598809 and its metabolite GSK685249: AUC (0-∞), Cmax, tmax, t½. | Pre-dose to 48h post dose.
Pair-wise correlation of BOLD signal changes in different image voxels and between selected brain structures during the alcohol-related cue paradigm and the Monetary Incentive Delay task, and in the brain resting state. | 1.5h (± 0.5h) after each dose (2 doses)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline